CLINICAL TRIAL: NCT05965518
Title: A Pilot Trial of High-Intensity Exercise to Combat Vascular and Cognitive Dysfunction in Older Adults With HIV
Brief Title: High-Intensity Exercise to Combat Vascular and Cognitive Dysfunction in Adults With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Raymond Jones, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300011502
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: HIV; Arterial Stiffness; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to high-intensity interval training or continuous moderate exercise for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity Interval Training (Experimental)
  Interventions: Behavioral: High-Intensity Interval Training
- Continuous Moderate Exercise (Active Comparator)
  Interventions: Behavioral: Continuous Moderate Exercise

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Following a 5-minute warm-up at 50% VO2peak, high and moderate-intensity exercise bouts alternate, progressing to five bouts of 4-minute high-intensity exercise (90% VO2peak), alternating with four 3-minute bouts of moderate-intensity exercise (50% VO2peak) by week 8, followed by a 5 minute cool-down. The total exercise time is 42 minutes.
  Arms: High-Intensity Interval Training
Behavioral: Continuous Moderate Exercise — Following a 4 minute warm-up at 50% VO2peak, the participant walks for up to 42 continuous minutes at 60% VO2peak, followed by a 4 minute cool-down. The total exercise time is 50 minutes.
  Arms: Continuous Moderate Exercise

SUMMARY:
This is a single site, randomized exercise trial with individuals at least 50 years of age living with HIV who experience suboptimal cognition. The overall goals of this proposal are to determine whether 16 weeks of structured high-intensity interval training (HIIT) can overcome vascular and cognitive impairments (Aim 1) to a greater extent than continuous moderate exercise. Additionally, investigator will seek to identify barriers to engagement in exercise and the participants' perceptions of the study and exercise interventions (Aim 2). This study will enroll 60 participants in Birmingham, Alabama. Data collection will occur at each visit, with baseline data collected at the initial visit with a 3-month follow-up occurring following completion of the intervention.

DETAILED DESCRIPTION:
This is a single site, randomized exercise trial with individuals at least 50 years of age living with HIV who experience suboptimal cognition. The overall goals of this proposal are to determine whether 12 weeks of structured high-intensity interval training (HIIT) can overcome vascular and cognitive impairments (Aim 1) to a greater extent than continuous moderate exercise. Additionally, investigator will seek to identify barriers to engagement in exercise and the participants' perceptions of the study and exercise interventions (Aim 2). This study will enroll 60 participants in Birmingham, Alabama.

Vascular function will be measured using pulse wave velocity. Cognition will be assessed using the full neuropsychological battery. Additionally, perceptions of exercise and the study as well as barriers to engaging in exercise will be determined through the analysis qualitative interviews.

The overall hypothesis is that HIIT will result in greater enhancements in vascular and cognitive function. The investigators expect that individuals randomized to HIIT will result in greater satisfaction with the protocol. Based on the data collected, the investigators seek to develop tailored intervention to promote successful aging among older people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older
* Sedentary lifestyle, deﬁned as < 150 min/wk moderate physical activity as assessed by CHAMPS questionnaire
* Neurocognitive Impairment (as assessed using the BRACE+
* Prescribed HIV ART for ≥ 12 months, with no current use of older drugs with established mitochondrial toxicity
* Able to speak, read, and write in English
* Willingness to participate in all study procedures

Exclusion Criteria:

* Diagnosis of mitochondrial disease
* Active substance abuse or factors preventing compliance or safety
* Uncontrolled hypertension, deﬁned as resting BP > 150/90 mmHG
* Chronic kidney disease
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically signiﬁcant aortic stenosis, history of cardiac arrest, use of a cardiac deﬁbrillator, or uncontrolled angina
* Acute myocardial infarction identiﬁed by medical history and ECG
* Pulmonary disease requiring the use of supplemental oxygen
* Poorly controlled diabetes
* Neuropsychologically Intact
* Orthopedic problems that limit ability to perform exercise
* Simultaneous participation in another intervention trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in vascular function | Baseline, Up to 16 weeks, 3-months Post-Intervention
  Arterial stiffness is a continuous measure of cardiovascular disease risk.
Change in cognitive function | Baseline, Up to 16 weeks, 3-months Post-Intervention
  Cognitive function will be measured using BRACE+, a neuropsychological battery

SECONDARY OUTCOMES:
Barriers to Engagement in Exercise | Baseline
  This will be assessed during qualitative interviews grounded in the Theoretical Domains Framework.
Perceptions of the Study and Exercise Interventions | Up to 16 weeks
  This will be assessed during qualitative interviews grounded in the Theoretical Domains Framework.

OTHER OUTCOMES:
Participant Safety, Adherence to the Intervention, Retention | Through study completion, an average of 6 months
  Participant safety will be assessed based on the number of adverse events which leads to termination of the exercise training. This will be registered as a binary outcome (yes/no). Adherence to the intervention will be measured based on the percentage of the exercise sessions that the participants attend. Retention at assessments will be measured by trial condition for each primary outcome assessment (e.g., immediately post-intervention and 3-months post-intervention). Participants will be considered retained if they complete the assessment visit in its entirety. It will be expressed as a percentage of participants with available outcome assessments immediately post-intervention and 3-months post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Jones, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant-level deidentified data will be preserved through deposition of the data in a controlled public repository. All aggregate datasets that can be shared publicly will be deposited in the NIH/NIA Repository, National Archive of Computerized Data on Aging (NACDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available no later than the time of an associated publication or end of the funding period, whichever comes first. NACDA guarantees data will be made available for ≥10 years
Access Criteria: De-identified individual participant data will be deposited into NACDA as restricted, which limits access to the data to qualified investigators with who must sign a data use agreement. NACDA requires users to submit a data use agreement. NACDA will review the data request for completeness and determine if an IRB approval is needed. Anyone who has submitted an approved data request and signed data use agreement on NACDA will be given access to the data without cost, for a set period.

REFERENCES:
- [Derived] Jones R, Hankes MJ, Vickers JK, Kulik GL, Jankowski CM, Oliveira V, Khuu V, Cook PF, Li P, Vance DE, Ivankova NV, Erlandson KM, Webel AR, Buford TW, Fazeli PL. Examining High-Intensity Exercise on Cognitive and Vascular Outcomes in Older Adults Living With HIV-A Research Protocol: Design and Rationale From Two Harmonized Clinical Studies in the Deep South. J Assoc Nurses AIDS Care. 2026 Jan-Feb 01;37(1):118-132. doi: 10.1097/JNC.0000000000000591. Epub 2025 Oct 1. PMID 41026763